CLINICAL TRIAL: NCT00079170
Title: A Pilot Study to Evaluate the Influence of Garlic on the Pharmacokinetics of Docetaxel in Patients With Metastatic Breast Cancer
Brief Title: Docetaxel Plus Garlic in Treating Patients With Locally Advanced or Metastatic Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000355083; NCI-04-C-0084; NCT00076193 (obsolete NCT alias)
Record Dates: First submitted 2004-03-08; First posted 2004-03-10 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2006-10

CONDITIONS: Breast Cancer
Keywords: male breast cancer; recurrent breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Docetaxel

INTERVENTIONS:
Dietary Supplement: garlic
Drug: docetaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, work in different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known whether garlic supplements affect the ability of docetaxel to kill tumor cells.

PURPOSE: This clinical trial is studying how well giving docetaxel together with garlic works in treating patients with locally advanced or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the clinical pharmacokinetic behavior of docetaxel with and without garlic tablets in patients with locally advanced or metastatic breast cancer.
* Determine the toxicity of this regimen in these patients.

Secondary

* Determine the incidence of enzyme and transporter polymorphism in patients treated with this regimen.

OUTLINE: This is a pilot, open-label study.

Patients receive docetaxel IV over 60 minutes on days 1, 8, and 15. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity. On days 5-17 of course 1, patients receive oral garlic twice daily. Patients have the option of continuing garlic tablets as long as they remain on study.

PROJECTED ACCRUAL: A total of 9-12 patients will be accrued for this study within 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the breast
* Incurable, locally advanced or metastatic disease for which therapy with docetaxel is a reasonable option
* No documentation of progressive disease while on docetaxel within the past 2 months
* Brain and/or leptomeningeal metastases are allowed only if all of the following criteria are met:

  * Asymptomatic on neurological examination, including after definitive radiotherapy
  * No corticosteroid therapy to control symptoms
  * Stable lesions
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Male or female

Menopausal Status

* Not specified

Performance status

* ECOG 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* Neutrophil count ≥ 1,200/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin normal
* ALT and AST ≤ 2 times ULN (3 times ULN with liver metastases)

Renal

* Creatinine normal OR
* Creatinine clearance ≥ 60 mL/min

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmias

Gastrointestinal

* No known gastric emptying disorders
* No persistent diarrhea

Other

* No uncontrolled diabetes mellitus
* No active infection
* No prior grade 3 or 4 allergic reaction attributed to compounds of similar biological composition to garlic, docetaxel, or Tween 80
* No other concurrent uncontrolled medical condition that would preclude study participation
* No psychiatric illness or social situation that would preclude study compliance
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception
* Must be able to ingest oral medication
* Lactic dehydrogenase ≤ 2 times ULN

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 3 weeks since prior immunotherapy
* No concurrent immunotherapy

  * Trastuzumab (Herceptin®) allowed after the first course of therapy at the discretion of the primary physician
* No concurrent pegfilgrastim

Chemotherapy

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* No other concurrent chemotherapy

Endocrine therapy

* See Disease Characteristics
* At least 2 weeks since prior hormonal therapy
* No concurrent hormonal therapy
* No concurrent megestrol during the first course of study treatment

Radiotherapy

* See Disease Characteristics
* At least 3 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery

* Not specified

Other

* More than 30 days (or 5 half-lives) since prior investigational therapy
* No concurrent aprepitant (Emend®)
* No concurrent or oral tetrahydrocannabinol (Marinol®) during the first course of study treatment
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational or anticancer medications
* No concurrent antiepileptic therapy
* No concurrent immunosuppressants
* No other concurrent herbal therapies during the first month of study participation
* No concurrent grapefruit juice during the first month of study participation
* No concurrent administration of the following:

  * Alprazolam
  * Cyclosporine
  * Diltiazem
  * Dofetilide
  * Erythromycin
  * Fluvoxamine
  * Itraconazole
  * Ketoconazole
  * Quinine
  * Hypericum perforatum (St. John's wort)
  * Tacrolimus
  * Theophylline
  * Warfarin
  * Zolpidem

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-01; Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael C. Cox, PharmD, Study Chair — NCI - Medical Oncology Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States